CLINICAL TRIAL: NCT03288571
Title: The Safety of Intra-parenchymal Wharton Jelly Mesenchymal Stem Cell Injection in the Treatment of Diabetic Nephropathy
Brief Title: Use of Wharton Jelly in Diabetic Nephropathy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sophia Al-Adwan (Other)
Collaborators: Jordan University of Science and Technology (Other); An-Najah National University (Other)
Responsible Party: Sponsor-Investigator, Sophia Al-Adwan, Clinical Co-ordinator, University of Jordan
Organization: University of Jordan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNJUCTC
Record Dates: First submitted 2017-08-08; First posted 2017-09-20 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Nephropathies
Keywords: Diabetes; nephropathy; Kidney; parenchyma; Wharton Jelly; Mesenchymal stem cells
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wharton Jelly Mesenchymal stem cells (Experimental): Intervention: Wharton Jelly Mesenchymal stem cells Site: Renal parenchyma Route of administration: ultrasound guided- intra-parenchymal total of 3 sites in each kidney.
  Number of doses: 3 doses 2 weeks apart for each kidney. Time interval between each dose: 2 weeks Total volume of cell suspension infused: 3 ml/kidney; each site will receive a 1 ml cell suspension with a total volume of 3 ml in each kidney.
  Interventions: Biological: Wharton Jelly Mesenchymal stem cells

INTERVENTIONS:
Biological: Wharton Jelly Mesenchymal stem cells — Wharton Jelly Mesenchymal stem cells will be injected in the renal parenchyma

SUMMARY:
Wharton Jelly derived Mesenchymal stem cells will be injected in the renal parenchyma of patients with Diabetic Nephropathy

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSCs) are to be isolated from Umbilical cord Wharton's Jelly obtained after normal full term delivery.

Samples will be tested for any bacterial or fungal growth as well as endotoxin and mycoplasma. The specific markers for MSCs identification will be analyzed by flow cytometry.

Cell suspension will then be injected in the renal parenchyma of patients diagnosed with diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Type 2 diabetes mellitus (DM) for ≥ 3 years.
* Estimated GFR (eGFR) 15-45 ml/min/1.73 m2 by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation on 2 or more consecutive measurements at least 30 days apart within the past 6 months, confirmed by isotope kidney scan.
* Urine protein-to-creatinine ratio (UPCR) ≥ 500 mg/mmol (in spot urine or in 24 hour urine collection) confirmed twice over a period of 6 months.
* Ultrasonographic kidney measurements ≥ 10 cm (for both kidneys).

Exclusion Criteria:

* Patients with uncontrolled hyper or hypo tension; (systolic pressure >160, <100: diastolic pressure < 60, >100) on two different occasions.
* Poor diabetic control: Hemoglobin A1c (HbA1c) > 10%.
* New use of hypoglycemic, antihypertensive and/or lipid lowering agent within the past 6 months.
* Increase in the dose of anti-hypertensive and/or hypoglycemic agent of the previous dose within the past 3 months.
* Current fasting total cholesterol >300 mg/dl.
* Current fasting total triglycerides >400 mg/dl.
* History of any cardiovascular events in the past 6 months.
* Pregnancy or lactating.
* Positive screening test for infectious diseases as per baseline work up.
* History of kidney transplant
* Systemic autoimmune disease.
* Receiving immunosuppressant medications.
* Patients with glomerulonephritis or any non-DM related kidney disease.
* Patients with any coagulation disorder.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 6 months
  * Number, frequency and severity of injection associated adverse events.
  * The nephrologist will record any adverse event at each follow up visit in addition to evaluation of the overall condition of the patient.

SECONDARY OUTCOMES:
Evaluation of the preliminary efficacy of the injection on kidney's Estimated Glomerular filtration rate | 12 months
  • Any positive changes in the patient's kidney function in terms of Estimated Gomerular filtration rate (mL/min/1.73 m²)
Evaluation of the preliminary efficacy of the injection on kidney's protein to creatinine ratio | 12 months
  Any positive changes in the patient's kidney function in terms of Urine protein to creatinine ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Abdalla Awidi, MD, Study Director — Cell Therapy Center

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: within one month of publication